CLINICAL TRIAL: NCT04847141
Title: A Multicenter, Randomized, Double-blind, Parallel Group Study to Evaluate the Safety and Efficacy of Anti-COVID-19 Immune Globulin (Human) 20% (C19-IG 20%) Versus Placebo in Asymptomatic Ambulatory Outpatients With Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection
Brief Title: A Study to Evaluate the Safety and Efficacy of C19-IG 20% in SARS-CoV-2 Infected Asymptomatic Ambulatory Outpatients
Acronym: COVID-19
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study Stopped for Futility
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GC2010; 2021-000269-34 (EudraCT Number)
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Results first posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: COVID-19; Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection
Keywords: Coronavirus disease; Severe acute respiratory syndrome coronavirus 2; SARS-CoV-2; COVID-19; Asymptomatic
MeSH Terms: conditions — COVID-19; Infections | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- C19-IG 20% 1 g (Experimental): Participants will receive 1 gram (g) of C19-IG 20% subcutaneous (SC) infusion containing one syringe of 5 milliliters (mL) C19-IG 20% plus one syringe of 5 mL sterile 0.9% sodium chloride (NaCl) on Day 1.
  Interventions: Biological: C19-IG 20%; Drug: 0.9% Sodium chloride
- C19-IG 20% 2 g (Experimental): Participants will receive 2 g of C19-IG 20% SC infusion containing two syringes 5 mL each of C19-IG 20% on Day 1.
  Interventions: Biological: C19-IG 20%
- Placebo (Placebo Comparator): Participants will receive C19-IG 20% matching placebo as SC infusion containing two syringes of 5 mL each sterile 0.9% NaCl injection on Day 1.
  Interventions: Drug: 0.9% Sodium chloride

INTERVENTIONS:
Biological: C19-IG 20% — Anti-COVID-19 Immune Globulin (Human) 20%
  Arms: C19-IG 20% 1 g; C19-IG 20% 2 g
Drug: 0.9% Sodium chloride — C19-IG 20% matching placebo
  Arms: C19-IG 20% 1 g; Placebo

SUMMARY:
The purpose of the study is to compare the efficacy of anti-COVID-19 immune globulin (human) 20% (C19-IG 20%) (2 doses) versus placebo with regard to the percentage of asymptomatic participants who remain asymptomatic, i.e., who do not develop symptomatic coronavirus disease 2019 (COVID-19) through Day 14 as per the protocol defined criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory male or female outpatients ≥ 18 years of age who have laboratory-confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection as determined by qualitative PCR (reverse transcriptase (RT)-PCR), or other commercial or public health assay approved by regulatory authorities as a diagnostic test for COVID-19 (inclusive of SARS-CoV-2 antigen testing or other approved rapid testing platforms) in any specimen ≤ 5 days prior to randomized treatment.
2. Asymptomatic with no constitutional COVID-19 illness (evident symptoms), specifically no fever, cough, shortness of breath, fatigue, anorexia, vomiting/diarrhea, headache that is unrelated to pre-existing conditions (example, migraine), sore throat that is unrelated to other pre-existing medical conditions (example, allergies, gastroesophageal reflux disease), myalgias, olfactory disorders unrelated with previous medical condition, or evidence of pneumonia at Screening.
3. Pulse oximetry peripheral oxygen saturation (SpO2) (oxygen saturation) on room air > 94% (i.e., 95% to 100%) at Screening.
4. National Early Warning Score (NEWS) ≤ 2 points at Screening.
5. Participant provides informed consent (ICF) prior to initiation of any study procedures.

Exclusion Criteria:

1. Participants who are admitted to hospital or for whom hospital admission is being planned at the time of Screening.
2. Participants requiring any form of oxygen supplementation at Screening.
3. Concurrent or planned treatment with other agents with actual or possible direct antiviral activity against SARS-CoV-2 including remdesivir.
4. Prior, concurrent or planned treatment with monoclonal antibodies (mAbs) against SARS-CoV-2
5. Have participated in a previous SARS-CoV-2 vaccine study OR outside of a study have received any SARS-CoV-2 vaccine of any kind.
6. Have a history of convalescent COVID-19 plasma treatment at Screening.
7. Fever (temperature ≥38.0° C [≥100.4° F]), measured orally, requirement for antipyretics to reduce temperature (administered for fever), and/or respiratory symptoms (cough, dyspnea) at Screening.
8. Clinical evidence of any significant acute or chronic disease that, in the opinion of the investigator, may place the participant at undue medical risk for study treatment.
9. The participant has had a known (documented) history of serious anaphylactic reaction to blood, any blood-derived plasma product or commercial immunoglobulin, or has known selective immunoglobulin A (IgA) deficiency with anti-IgA antibodies.
10. Decompensated congestive heart failure or renal failure with fluid overload. This includes currently uncontrolled congestive heart failure New York Heart Association Class III or IV stage heart failure.
11. Participants for whom there is limitation of therapeutic effort such as "Do not resuscitate" status.
12. Currently participating in another interventional clinical trial with investigational medical product or device.
13. Participants with known (documented) thrombotic complications to polyclonal intravenous immune globulin (IVIG) therapy in the past.
14. Participant has medical condition (other than COVID-19) that is projected to limit lifespan to ≤ 1 year.
15. Participant has history of drug or alcohol abuse within the past 12 months.
16. Participant is unwilling to commit to follow-up visits.
17. Women who are pregnant or breastfeeding, or if of childbearing potential, unwilling to practice a highly effective method of contraception (oral, injectable, or implanted hormonal methods of contraception, placement of an intrauterine device or intrauterine system, condom, or occlusive cap with spermicidal foam/gel/cream/suppository, male sterilization, or true abstinence) throughout the study.

    * True abstinence: When this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods], declaration of abstinence for the duration of a trial, and withdrawal are not acceptable methods of contraception).
    * Note: Women who are >55 years and with the absence of menses in the last 12 months are considered to be not of childbearing potential. Female participants of childbearing potential must have a negative test for pregnancy blood or urine human chorionic gonadotropin (hCG)-based assay at Screening/Baseline Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oriol Mitjà, MD, Principal Investigator — omitja@lluita.org, +3493 4978339
Locations (12):
- Spain (12):
  - CAP Gornal, L'Hospitalet de Llobregat, Barcelona
  - CAP Navàs, Navàs, Barcelona
  - CAP Sant Fèlix, Sabadell, Barcelona
  - Centro de Salud Nuestra Señora del Pilar, Alcalá de Henares, Madrid
  - Centro de Salud Presentación Sabio, Móstoles, Madrid
  - CAP Manso, Barcelona
  - CAP Maluquer Salvador, Girona
  - Centro de Salud San Andrés, Madrid
  - Centro de Salud Fuentelarreina, Madrid
  - Centro de Salud Hacienda de Pavones Sureste, Madrid
  - Centro de Salud Isla de Oza Noroeste, Madrid
  - Hospital Sant Pau i Santa Tecla, Tarragona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alemany A, Millat-Martinez P, Corbacho-Monne M, Suner C, Galvan-Casas C, Carrera C, Ouchi D, Prat N, Ara J, Nadal N, Riel R, Funollet B, Ojeda-Ciurana C, Balague LE, Salvador-Gonzalez B, Arcarons AF, Vidal-Alaball J, Del Cura-Gonzalez MI, Barrientos RR, Ramos-Blanes R, Bou AA, Mondou E, Torres M, Campins N, Sanz A, Tang Y, Rodriguez-Arias MA, Bassat Q, Clotet B; GC2010 STUDY GROUP; Mitja O. Subcutaneous anti-COVID-19 hyperimmune immunoglobulin for prevention of disease in asymptomatic individuals with SARS-CoV-2 infection: a double-blind, placebo-controlled, randomised clinical trial. EClinicalMedicine. 2023 Mar 10;57:101898. doi: 10.1016/j.eclinm.2023.101898. eCollection 2023 Mar. PMID 36936402

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at 5 centers in Spain. The study was conducted from 28 April 2021 to 27 December 2021.
Pre-assignment Details: Participants with Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-Cov-2) infection were randomized in 1:1:1 ratio to receive anti-COVID-19 Immune Globulin (Human) 20% [C19-IG 20%] 1 gram (g), C19-IG 20% 2 g, and placebo. A total of 555 participants were screened and 465 participants were randomized in the study. Among these, 461 participants were dosed, and 430 participants completed the study.
Groups:
- C19-IG 20% 1 g: Participants received 1 g of C19-IG 20% SC infusion containing one syringe of 5 mL C19-IG 20% plus one syringe of 5 mL sterile 0.9% NaCl on Day 1.
- C19-IG 20% 2 g: Participants received 2 g of C19-IG 20% SC infusion containing two syringes 5 mL each of C19-IG 20% on Day 1.
- Placebo: Participants received C19-IG 20% matching placebo as SC infusion containing two syringes of 5 mL each sterile 0.9% NaCl injection on Day 1.
Period: Overall Study
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Started (Started participants were defined as participants who were also dosed.) | 152 | 153 | 156
Completed | 142 | 143 | 145
Not Completed | 10 | 10 | 11
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 4 | 3
Not completed — Lost to Follow-up | 7 | 5 | 7
Not completed — Reason not Specified | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized. Modified ITT (mITT) population included the subset of ITT participants who were also dosed.
Groups:
- Total: Total of all reporting groups
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo | Total
Number analyzed (Participants) | 152 | 153 | 156 | 461
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (12.76) | 41.1 (12.40) | 38.8 (13.33) | 39.6 (12.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 62 | 69 | 197
  Male | 86 | 91 | 87 | 264
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 32 | 45 | 117
  Not Hispanic or Latino | 112 | 121 | 111 | 344
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 4 | 6 | 3 | 13
  White | 138 | 140 | 140 | 418
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 9 | 6 | 9 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Asymptomatic Participants Who Remained Asymptomatic, i.e., Who Did Not Develop Symptomatic COVID-19 Through Day 14
Description: Participants were described as symptomatic if they a. experienced at least two of the following systemic symptoms: fever (≥38 ºC), chills, myalgia, headache, sore throat, cough, fatigue that interferes with activities of daily living, new olfactory/taste disorder(s), and vomiting/diarrhea, b. experienced at least one of the following respiratory signs/symptoms: new or worsening shortness of breath or difficulty breathing; c. experienced a peripheral oxygen saturation by pulse oximetry (SpO2) <94% on room air; or d. had radiographical evidence of pneumonia. The percentage of participants who meet the primary endpoint within each treatment group was presented along with a two-sided exact (Clopper-Pearson) 95% confidence interval (CI).
Time Frame: Up to Day 14
Population: mITT population included the subset of ITT participants (all randomized participants) who were also dosed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 152 | 153 | 156
percentage of participants | 59.9 [51.6 to 67.7] | 64.7 [56.6 to 72.3] | 63.5 [55.4 to 71.0]
Statistical Analysis 1: Comparison: C19-IG 20% 1 g vs Placebo; Test type: Superiority; p = 0.5167, Chi-squared — p-value was calculated using Chi-square test with 5% level of significance to test the null hypothesis of no difference in the percentage of participants meeting the primary efficacy endpoint between C19-IG 20% 1 g and placebo; Difference in Percentage = -3.6, 95% CI 2-sided [-14.6 to 7.4] — 95% CI for percentage difference between C19-IG 20% 1 g dose group and placebo was calculated using the exact unconditional method
Statistical Analysis 2: Comparison: C19-IG 20% 2 g vs Placebo; Test type: Superiority; p = 0.8197, Chi-squared — p-value was calculated using Chi-square test with 5% level of significance to test the null hypothesis of no difference in the percentage of participants meeting the primary efficacy endpoint between C19-IG 20% 2 g and placebo; Difference in Percentage = 1.2, 95% CI 2-sided [-9.6 to 12.0] — 95% CI for percentage difference between C19-IG 20% 2 g dose group and placebo was calculated using the exact unconditional method

2. Secondary Outcome: Change From Baseline in SARS-CoV-2 Viral Load (log10 Copies/mL)
Description: Mean change from baseline (CFB) in log10 SARS-CoV-2 viral load at Days 7 and 14 was assessed.
Time Frame: Baseline to Day 7 and Day 14
Population: mITT population included the subset of ITT participants who were also dosed. Here, "Number analyzed" is the number of participants with data available for analysis at the given time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 copies/mL
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 152 | 153 | 156
log10 copies/mL
  Change from Baseline at Day 7: number analyzed (Participants) | 143 | 140 | 147
  Change from Baseline at Day 7 | -1.49 [-1.74 to -1.25] | -1.76 [-2.01 to -1.51] | -1.59 [-1.83 to -1.35]
  Change from Baseline at Day 14: number analyzed (Participants) | 135 | 134 | 137
  Change from Baseline at Day 14 | -2.80 [-2.97 to -2.64] | -3.02 [-3.19 to -2.85] | -2.91 [-3.08 to -2.75]
Statistical Analysis 1: Comparison: C19-IG 20% 1 g vs Placebo; Day 7; Test type: Superiority; p = 0.5756, ANCOVA; Least squares (LS) Mean Difference = 0.10, 95% CI 2-sided [-0.24 to 0.44] — 95% CI for the difference in LS Mean between 1 g C19-IG 20% dose group & placebo was calculated using ANCOVA model, including CFB value as dependent variable; treatment group as fixed effect; & baseline viral load value, age, & gender as covariates
Statistical Analysis 2: Comparison: C19-IG 20% 2 g vs Placebo; Day 7; Test type: Superiority; p = 0.3289, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.52 to 0.17] — 95% CI for the difference in LS Mean between 2 g C19-IG 20% dose group & placebo was calculated using ANCOVA model, including CFB value as dependent variable; treatment group as fixed effect; & baseline viral load value, age, & gender as covariates
Statistical Analysis 3: Comparison: C19-IG 20% 1 g vs Placebo; Day 14; Test type: Superiority; p = 0.3418, ANCOVA; LS Mean Difference = 0.11, 95% CI 2-sided [-0.12 to 0.34] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: C19-IG 20% 2 g vs Placebo; Day 14; Test type: Superiority; p = 0.3688, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.34 to 0.13] — [estimate comment as in outcome 2, analysis 2]

3. Secondary Outcome: Percentage of Participants Who Remained in an Outpatient Setting and Maintained SpO2 ≥94% on Room Air on Day 3, Day 7, and Day 14
Description: An outpatient setting was defined as no hospitalization or intensive care unit (ICU) admission through Days 3, 7, and 14. The percentage of participants who remained in an outpatient setting and maintained SpO2 ≥94% on room air at each timepoint within each treatment group were presented along with a two-sided exact (Clopper-Pearson) 95% CI. p-value and 95% CI were not estimable for C19-IG 20% 1 g vs placebo as all participants had remained in an outpatient setting and maintained SpO2 ≥94% on Room Air in C19-IG 20% 1 g and placebo arm on Day 3.
Time Frame: Day 3, Day 7, and Day 14
Population: mITT population included the subset of ITT participants who were also dosed. Here, "Number analyzed" is number of participants with data available for analysis at given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 152 | 153 | 156
percentage of participants
  Day 3: number analyzed (Participants) | 151 | 152 | 156
  Day 3 | 100 [97.6 to 100] | 98.7 [95.3 to 99.8] | 100 [97.7 to 100]
  Day 7: number analyzed (Participants) | 149 | 151 | 156
  Day 7 | 100 [97.6 to 100] | 96.7 [92.4 to 98.9] | 98.7 [95.5 to 99.8]
  Day 14: number analyzed (Participants) | 148 | 149 | 154
  Day 14 | 95.3 [90.5 to 98.1] | 94.0 [88.8 to 97.2] | 96.1 [91.7 to 98.6]
Statistical Analysis 1: Comparison: C19-IG 20% 2 g vs Placebo; Day 3; Test type: Superiority; p = 0.1506, Chi-squared — p-value was calculated using Chi-square test with 5% level of significance to test the null hypothesis of no difference in the percentage of participants who remained in an outpatient setting & maintained SpO2≥94% between C19-IG 20% 2 g & placebo; Difference in Percentage = -1.3, 95% CI 2-sided [-4.7 to 1.2] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: C19-IG 20% 1 g vs Placebo; Day 7; Test type: Superiority; p = 0.1655, Chi-squared — p-value was calculated using Chi-square test with 5% level of significance to test the null hypothesis of no difference in the percentage of participants who remained in an outpatient setting & maintained SpO2≥94% between C19-IG 20% 1 g & placebo; Difference in Percentage = 1.3, 95% CI 2-sided [-1.3 to 4.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: C19-IG 20% 2 g vs Placebo; Day 7; Test type: Superiority; p = 0.2337, Chi-squared — [p-value comment as in outcome 3, analysis 1]; Difference in Percentage = -2.0, 95% CI 2-sided [-6.5 to 1.7] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: C19-IG 20% 1 g vs Placebo; Day 14; Test type: Superiority; p = 0.7212, Chi-squared — [p-value comment as in outcome 3, analysis 2]; Difference in Percentage = -0.8, 95% CI 2-sided [-6.1 to 4.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: C19-IG 20% 2 g vs Placebo; Day 14; Test type: Superiority; p = 0.3897, Chi-squared — [p-value comment as in outcome 3, analysis 1]; Difference in Percentage = -2.1, 95% CI 2-sided [-7.8 to 3.1] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Percentage of Participants Negative for SARS-CoV-2 by Polymerase Chain Reaction (PCR) Test at Multiple Timepoints Through Day 14 and Through Day 29
Description: The percentage of participants with negative SARS-CoV-2 by PCR through Day 14 and Day 29 within each treatment group was presented along with a two-sided exact (Clopper-Pearson) 95% CI.
Time Frame: Day 3, Day 7, Day 14, and Day 29
Population: mITT population included the subset of ITT participants who were also dosed. Here, "Number analyzed" is the number of participants with non-missing test results at the given visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 152 | 153 | 156
percentage of participants
  Day 3: number analyzed (Participants) | 148 | 148 | 154
  Day 3 | 29.1 [21.9 to 37.1] | 30.4 [23.1 to 38.5] | 26.0 [19.3 to 33.7]
  Day 7: number analyzed (Participants) | 143 | 141 | 147
  Day 7 | 37.8 [29.8 to 46.3] | 44.0 [35.6 to 52.6] | 36.1 [28.3 to 44.4]
  Day 14: number analyzed (Participants) | 135 | 135 | 137
  Day 14 | 65.2 [56.5 to 73.2] | 74.1 [65.8 to 81.2] | 67.2 [58.6 to 74.9]
  Day 29: number analyzed (Participants) | 125 | 127 | 124
  Day 29 | 92.0 [85.8 to 96.1] | 89.0 [82.2 to 93.8] | 87.1 [79.9 to 92.4]
Statistical Analysis 1: Comparison: C19-IG 20% 1 g vs Placebo; Day 3; Test type: Superiority; p = 0.5489, Chi-squared — p-value was calculated using Chi-square test with 5% level of significance to test the null hypothesis of no difference in the percentage of participants who had a negative test result between C19-IG 20% 1 g dose group and placebo; Difference in Percentage = 3.1, 95% CI 2-sided [-7.1 to 13.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: C19-IG 20% 2 g vs Placebo; Day 3; Test type: Superiority; p = 0.3920, Chi-squared — p-value was calculated using Chi-square test with 5% level of significance to test the null hypothesis of no difference in the percentage of participants who had a negative test result between C19-IG 20% 2 g dose group and placebo; Difference in Percentage = 4.4, 95% CI 2-sided [-5.8 to 14.7] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: C19-IG 20% 1 g vs Placebo; Day 7; Test type: Superiority; p = 0.7632, Chi-squared — [p-value comment as in outcome 4, analysis 1]; Difference in Percentage = 1.7, 95% CI 2-sided [-9.5 to 12.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: C19-IG 20% 2 g vs Placebo; Day 7; Test type: Superiority; p = 0.1702, Chi-squared — [p-value comment as in outcome 4, analysis 2]; Difference in Percentage = 7.9, 95% CI 2-sided [-3.6 to 19.2] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: C19-IG 20% 1 g vs Placebo; Day 14; Test type: Superiority; p = 0.7316, Chi-squared — [p-value comment as in outcome 4, analysis 1]; Difference in Percentage = -2.0, 95% CI 2-sided [-13.3 to 9.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: C19-IG 20% 2 g vs Placebo; Day 14; Test type: Superiority; p = 0.2104, Chi-squared — [p-value comment as in outcome 4, analysis 2]; Difference in Percentage = 6.9, 95% CI 2-sided [-4.2 to 18.0] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: C19-IG 20% 1 g vs Placebo; Day 29; Test type: Superiority; p = 0.2059, Chi-squared — [p-value comment as in outcome 4, analysis 1]; Difference in Percentage = 4.9, 95% CI 2-sided [-2.9 to 13.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: C19-IG 20% 2 g vs Placebo; Day 29; Test type: Superiority; p = 0.6463, Chi-squared — [p-value comment as in outcome 4, analysis 2]; Difference in Percentage = 1.9, 95% CI 2-sided [-6.5 to 10.3] — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: Time to Negative SARS-CoV-2 PCR From Baseline Through Day 29
Description: The first negative test result was defined as the first PCR negative result after the first PCR positive result. Kaplan-Meier method was used for analysis. Participants who did not have any viral load data or had negative test results through the study were excluded from the KM analysis.
Time Frame: Baseline to Day 29
Population: mITT population included the subset of ITT participants who were also dosed. Here, "Overall number of participants analyzed" is the participants who achieved negative test results through Day 29.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 101 | 95 | 112
days | 14 [14 to 15] | 14 [14 to 15] | 14 [14 to 15]
Statistical Analysis 1: Comparison: C19-IG 20% 1 g vs Placebo; Test type: Superiority; p = 0.9033, Log Rank
Statistical Analysis 2: Comparison: C19-IG 20% 2 g vs Placebo; Test type: Superiority; p = 0.5456, Log Rank

6. Secondary Outcome: Percentage of Participants Who Required Oxygen (O2) Supplementation on or Before Day 29
Description: The percentage of participants requiring oxygen supplementation through Day 29 within each treatment group was presented along with a two-sided exact (Clopper-Pearson) 95% CI.
Time Frame: Up to Day 29
Population: mITT population included the subset of ITT participants who were also dosed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 152 | 153 | 156
percentage of participants | 2.0 [0.4 to 5.7] | 3.9 [1.5 to 8.3] | 1.3 [0.2 to 4.6]
Statistical Analysis 1: Comparison: C19-IG 20% 1 g vs Placebo; Test type: Superiority; p = 0.6311, Chi-squared — p-value was calculated using Chi-square test with 5% level of significance to test the null hypothesis of no difference in the percentage of participants who required oxygen supplementation between C19-IG 20% 1 g dose group and placebo; Difference in Percentage = 0.79, 95% CI 2-sided [-2.9 to 4.6] — 95% CI for percentage difference between each of 1 g C19-IG 20% dose group and placebo was calculated using the exact unconditional method
Statistical Analysis 2: Comparison: C19-IG 20% 2 g vs Placebo; Test type: Superiority; p = 0.1441, Chi-squared — p-value was calculated using Chi-square test with 5% level of significance to test the null hypothesis of no difference in the percentage of participants who required oxygen supplementation between C19-IG 20% 2 g dose group and placebo; Difference in Percentage = 2.6, 95% CI 2-sided [-1.2 to 7.3] — 95% CI for percentage difference between each of 2 g C19-IG 20% dose group and placebo was calculated using the exact unconditional method

7. Secondary Outcome: Duration of Any Oxygen Use Through Day 29
Description: The duration (number of days) of any oxygen use from Day 1 through Day 29 was calculated based on the start/stop date of using oxygen supplementation.
Time Frame: Up to Day 29
Population: mITT population included the subset of ITT participants who were also dosed. Here, "Overall number of participants analyzed" is the number of participants who required oxygen supplementation.
Measure: Median (Full Range); unit: days
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 3 | 5 | 2
days | 7.0 [6 to 9] | 7.0 [2 to 8] | 9.5 [4 to 15]
Statistical Analysis 1: Comparison: C19-IG 20% 1 g vs Placebo; Test type: Superiority; p = 0.8555, ANCOVA; LS Mean (LSM) Difference = 0.02, 95% CI 2-sided [-0.23 to 0.27] — 95% CI for difference in LSM between 1 g C19-IG 20% & placebo was calculated using an ANCOVA model,with number of days on oxygen as dependent variable & treatment group as fixed effect,adjusting for baseline characteristics(including age & gender)
Statistical Analysis 2: Comparison: C19-IG 20% 2 g vs Placebo; Test type: Superiority; p = 0.8108, ANCOVA; LS Mean Difference = 0.03, 95% CI 2-sided [-0.22 to 0.28] — 95% CI for difference in LSM between 2 g C19-IG 20% & placebo was calculated using an ANCOVA model,with number of days on oxygen as dependent variable & treatment group as fixed effect,adjusting for baseline characteristics(including age & gender)

8. Secondary Outcome: Absolute Value Score on a 7-point Ordinal Scale
Description: The ordinal scale is a 7-point scale ranging from 1 to 7 used to measure clinical status of a participant based on the following points: 1) death; 2) hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) hospitalized, requiring supplemental oxygen; 5) hospitalized, not requiring supplemental oxygen; 6) not hospitalized, limitation on activities; and 7) not hospitalized, no limitations on activities. A higher score indicates less severity.
Time Frame: Baseline, Day 7, 14, and 29
Population: mITT population included the subset of ITT participants who were also dosed. Here, "Number analyzed" is the number of participants with data available at the given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 152 | 153 | 156
score on a scale
  Baseline | 7.0 (0.00) | 7.0 (0.08) | 7.0 (0.08)
  Day 7: number analyzed (Participants) | 148 | 147 | 154
  Day 7 | 7.0 (0.08) | 7.0 (0.16) | 7.0 (0.19)
  Day 14: number analyzed (Participants) | 146 | 148 | 146
  Day 14 | 7.0 (0.32) | 6.9 (0.48) | 7.0 (0.08)
  Day 29: number analyzed (Participants) | 142 | 144 | 145
  Day 29 | 7.0 (0.20) | 7.0 (0.14) | 7.0 (0.08)

9. Secondary Outcome: Mean Change From Baseline in the 7-point Ordinal Scale
Description: The ordinal scale is a 7-point scale ranging from 1 to 7 used to measure clinical status of a participant based on the following points: 1) death; 2) hospitalized, on invasive mechanical ventilation or ECMO; 3) hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) hospitalized, requiring supplemental oxygen; 5) hospitalized, not requiring supplemental oxygen; 6) not hospitalized, limitation on activities; and 7) not hospitalized, no limitations on activities. A higher score indicates less severity. The analysis was performed by using a linear mixed-effects model for repeated measures (MMRM).
Time Frame: Baseline to Day 7, Day 14, and Day 29
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 152 | 153 | 156
score on a scale
  Change from Baseline at Day 7: number analyzed (Participants) | 148 | 147 | 154
  Change from Baseline at Day 7 | -0.00 [-0.03 to 0.02] | -0.02 [-0.05 to 0.00] | -0.04 [-0.06 to -0.01]
  Change from Baseline at Day 14: number analyzed (Participants) | 146 | 148 | 146
  Change from Baseline at Day 14 | -0.05 [-0.11 to 0.00] | -0.07 [-0.12 to -0.01] | -0.00 [-0.06 to 0.05]
  Change from Baseline at Day 29: number analyzed (Participants) | 142 | 144 | 145
  Change from Baseline at Day 29 | -0.04 [-0.06 to -0.01] | -0.02 [-0.04 to 0.01] | -0.00 [-0.03 to 0.02]
Statistical Analysis 1: Comparison: C19-IG 20% 1 g vs Placebo; Day 7; Test type: Superiority; p = 0.0692, Kenward-Roger — p-value was calculated using restricted maximum likelihood with the Kenward-Roger method; LS Mean Difference = 0.03, 95% CI 2-sided [-0.00 to 0.07] — 95% CI for difference in LS Mean between C19-IG 20% 1 g dose group and placebo was calculated using restricted maximum likelihood with the Kenward-Roger method for calculating the denominator degrees of freedom
Statistical Analysis 2: Comparison: C19-IG 20% 2 g vs Placebo; Day 7; Test type: Superiority; p = 0.4956, Kenward-Roger — p-value was calculated using restricted maximum likelihood with the Kenward-Roger method; LS Mean Difference = 0.01, 95% CI 2-sided [-0.02 to 0.05] — 95% CI for difference in LS Mean between C19-IG 20% 2 g dose group and placebo was calculated using restricted maximum likelihood with the Kenward-Roger method for calculating the denominator degrees of freedom
Statistical Analysis 3: Comparison: C19-IG 20% 1 g vs Placebo; Day 14; Test type: Superiority; p = 0.2200, Kenward-Roger — p-value was calculated using restricted maximum likelihood with the Kenward-Roger method; LS Mean Difference = -0.05, 95% CI 2-sided [-0.13 to 0.03] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: C19-IG 20% 2 g vs Placebo; Day 14; Test type: Superiority; p = 0.0906, Kenward-Roger — p-value was calculated using restricted maximum likelihood with the Kenward-Roger method; LS Mean Difference = -0.07, 95% CI 2-sided [-0.14 to 0.01] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 5: Comparison: C19-IG 20% 1 g vs Placebo; Day 29; Test type: Superiority; p = 0.0439, Kenward-Roger — p-value was calculated using restricted maximum likelihood with the Kenward-Roger method; LS Mean Difference = -0.04, 95% CI 2-sided [-0.07 to -0.00] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: C19-IG 20% 2 g vs Placebo; Day 29; Test type: Superiority; p = 0.4128, Kenward-Roger — p-value was calculated using restricted maximum likelihood with the Kenward-Roger method; LS Mean Difference = -0.01, 95% CI 2-sided [-0.05 to 0.02] — [estimate comment as in outcome 9, analysis 2]

10. Secondary Outcome: Percentage of Participants in Each Severity Category of the 7-point Ordinal Scale
Description: The ordinal scale is a 7-point scale ranging from 1 to 7 used to measure clinical status of a participant based on the following points: 1) death; 2) hospitalized, on invasive mechanical ventilation or ECMO; 3) hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) hospitalized, requiring supplemental oxygen; 5) hospitalized, not requiring supplemental oxygen; 6) not hospitalized, limitation on activities; and 7) not hospitalized, no limitations on activities.
Time Frame: Days 1, 7, 14, and 29
Population: mITT population included the subset of ITT participants who were also dosed. Here, "Number analyzed" is the number of participants with data available at the given time point in each treatment group. The percentage values are rounded off to the nearest decimal point.
Measure: Number; unit: percentage of participants
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 152 | 153 | 156
percentage of participants
  Day 1: Death | 0.0 | 0.0 | 0.0
  Day 1: Hospitalized, on invasive mechanical ventilation/ ECMO | 0.0 | 0.0 | 0.0
  Day 1: Hospitalized, on non-invasive ventilation or high flow oxygen devices | 0.0 | 0.0 | 0.0
  Day 1: Hospitalized, requiring supplemental oxygen | 0.0 | 0.0 | 0.0
  Day 1: Hospitalized, not requiring supplemental oxygen | 0.0 | 0.0 | 0.0
  Day 1: Not hospitalized, limitation on activities | 0.0 | 0.7 | 0.6
  Day 1: Not hospitalized, no limitations on activities | 100 | 99.3 | 99.4
  Day 7: Death: number analyzed (Participants) | 148 | 147 | 154
  Day 7: Death | 0.0 | 0.0 | 0.0
  Day 7: Hospitalized, on invasive mechanical ventilation/ ECMO: number analyzed (Participants) | 148 | 147 | 154
  Day 7: Hospitalized, on invasive mechanical ventilation/ ECMO | 0.0 | 0.0 | 0.0
  Day 7: Hospitalized, on non-invasive ventilation or high flow oxygen devices: number analyzed (Participants) | 148 | 147 | 154
  Day 7: Hospitalized, on non-invasive ventilation or high flow oxygen devices | 0.0 | 0.0 | 0.0
  Day 7: Hospitalized, requiring supplemental oxygen: number analyzed (Participants) | 148 | 147 | 154
  Day 7: Hospitalized, requiring supplemental oxygen | 0.0 | 0.0 | 0.0
  Day 7: Hospitalized, not requiring supplemental oxygen: number analyzed (Participants) | 148 | 147 | 154
  Day 7: Hospitalized, not requiring supplemental oxygen | 0.0 | 0.0 | 0.0
  Day 7: Not hospitalized, limitation on activities: number analyzed (Participants) | 148 | 147 | 154
  Day 7: Not hospitalized, limitation on activities | 0.7 | 2.7 | 3.9
  Day 7: Not hospitalized, no limitations on activities: number analyzed (Participants) | 148 | 147 | 154
  Day 7: Not hospitalized, no limitations on activities | 99.3 | 97.3 | 96.1
  Day 14: Death: number analyzed (Participants) | 146 | 148 | 146
  Day 14: Death | 0.0 | 0.0 | 0.0
  Day 14: Hospitalized, on invasive mechanical ventilation/ ECMO: number analyzed (Participants) | 146 | 148 | 146
  Day 14: Hospitalized, on invasive mechanical ventilation/ ECMO | 0.0 | 0.0 | 0.0
  Day 14: Hospitalized, on non-invasive ventilation or high flow oxygen devices: number analyzed (Participants) | 146 | 148 | 146
  Day 14: Hospitalized, on non-invasive ventilation or high flow oxygen devices | 0.0 | 1.4 | 0.0
  Day 14: Hospitalized, requiring supplemental oxygen: number analyzed (Participants) | 146 | 148 | 146
  Day 14: Hospitalized, requiring supplemental oxygen | 0.7 | 0.0 | 0.0
  Day 14: Hospitalized, not requiring supplemental oxygen: number analyzed (Participants) | 146 | 148 | 146
  Day 14: Hospitalized, not requiring supplemental oxygen | 0.7 | 0.0 | 0.0
  Day 14: Not hospitalized, limitation on activities: number analyzed (Participants) | 146 | 148 | 146
  Day 14: Not hospitalized, limitation on activities | 1.4 | 2.0 | 0.7
  Day 14: Not hospitalized, no limitations on activities: number analyzed (Participants) | 146 | 148 | 146
  Day 14: Not hospitalized, no limitations on activities | 97.3 | 96.6 | 99.3
  Day 29: Death: number analyzed (Participants) | 142 | 144 | 145
  Day 29: Death | 0.0 | 0.0 | 0.0
  Day 29: Hospitalized, on invasive mechanical ventilation/ ECMO: number analyzed (Participants) | 142 | 144 | 145
  Day 29: Hospitalized, on invasive mechanical ventilation/ ECMO | 0.0 | 0.0 | 0.0
  Day 29: Hospitalized, on non-invasive ventilation or high flow oxygen devices: number analyzed (Participants) | 142 | 144 | 145
  Day 29: Hospitalized, on non-invasive ventilation or high flow oxygen devices | 0.0 | 0.0 | 0.0
  Day 29: Hospitalized, requiring supplemental oxygen: number analyzed (Participants) | 142 | 144 | 145
  Day 29: Hospitalized, requiring supplemental oxygen | 0.0 | 0.0 | 0.0
  Day 29: Hospitalized, not requiring supplemental oxygen: number analyzed (Participants) | 142 | 144 | 145
  Day 29: Hospitalized, not requiring supplemental oxygen | 0.0 | 0.0 | 0.0
  Day 29: Not hospitalized, limitation on activities: number analyzed (Participants) | 142 | 144 | 145
  Day 29: Not hospitalized, limitation on activities | 4.2 | 2.1 | 0.7
  Day 29: Not hospitalized, no limitations on activities: number analyzed (Participants) | 142 | 144 | 145
  Day 29: Not hospitalized, no limitations on activities | 95.8 | 97.9 | 99.3

11. Secondary Outcome: Change From Baseline in National Early Warning Score (NEWS)
Description: The NEWS has demonstrated an ability to classify participants at risk of poor outcomes. This score is based on 7 clinical parameters (respiration rate, oxygen saturation, any supplemental oxygen, temperature, systolic blood pressure (BP), heart rate, level of consciousness [Alert, Voice, Pain, Unresponsive]). A score of 0 to 3 was allocated to each parameter except supplemental oxygen use (score of 0 or 2) and level of consciousness (score of 0 [alert, normal health condition] or 3 [altered mental state/confusion, worst health condition]). All parameter scores were summed to get an aggregate NEWS assessment. Scoring for NEWS ranges from 0 to 20, with higher scores meaning more severity/higher clinical risk: low risk (score 1 to 4); medium risk (score 5 to 6); high risk (score 7 to 20). The analysis is performed by using a linear MMRM.
Time Frame: Baseline to Day 7, Day 14, and Day 29
Population: mITT population included the subset of ITT participants who were also dosed. Here, "Number analyzed" is the number of participants with a non-missing NEWS total score at the given time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 152 | 153 | 156
score on a scale
  Change from Baseline at Day 7: number analyzed (Participants) | 137 | 138 | 146
  Change from Baseline at Day 7 | 0.70 [0.50 to 0.90] | 0.78 [0.58 to 0.98] | 0.70 [0.51 to 0.90]
  Change from Baseline at Day 14: number analyzed (Participants) | 132 | 134 | 138
  Change from Baseline at Day 14 | 0.68 [0.49 to 0.87] | 0.65 [0.46 to 0.84] | 0.67 [0.48 to 0.86]
  Change from Baseline at Day 29: number analyzed (Participants) | 121 | 123 | 121
  Change from Baseline at Day 29 | 0.61 [0.43 to 0.79] | 0.59 [0.40 to 0.77] | 0.46 [0.27 to 0.64]
Statistical Analysis 1: Comparison: C19-IG 20% 1 g vs Placebo; Day 7; Test type: Superiority; p = 0.9713, Kenward-Roger — p-value was calculated using restricted maximum likelihood with the Kenward-Roger method; LS Mean Difference = -0.01, 95% CI 2-sided [-0.28 to 0.27] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: C19-IG 20% 2 g vs Placebo; Day 7; Test type: Superiority; p = 0.5985, Kenward-Roger — p-value was calculated using restricted maximum likelihood with the Kenward-Roger method; LS Mean Difference = 0.07, 95% CI 2-sided [-0.20 to 0.35] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 3: Comparison: C19-IG 20% 1 g vs Placebo; Day 14; Test type: Superiority; p = 0.9209, Kenward-Roger — p-value was calculated using restricted maximum likelihood with the Kenward-Roger method; LS Mean Difference = 0.01, 95% CI 2-sided [-0.25 to 0.28] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: C19-IG 20% 2 g vs Placebo; Day 14; Test type: Superiority; p = 0.9181, Kenward-Roger — p-value was calculated using restricted maximum likelihood with the Kenward-Roger method; LS Mean Difference = -0.01, 95% CI 2-sided [-0.28 to 0.25] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 5: Comparison: C19-IG 20% 1 g vs Placebo; Day 29; Test type: Superiority; p = 0.2443, Kenward-Roger — p-value was calculated using restricted maximum likelihood with the Kenward-Roger method; LS Mean Difference = 0.15, 95% CI 2-sided [-0.11 to 0.41] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: C19-IG 20% 2 g vs Placebo; Day 29; Test type: Superiority; p = 0.3233, Kenward-Roger — p-value was calculated using restricted maximum likelihood with the Kenward-Roger method; LS Mean Difference = 0.13, 95% CI 2-sided [-0.13 to 0.39] — [estimate comment as in outcome 9, analysis 2]

12. Secondary Outcome: Percentage of Participants Who Required At Least One COVID-19 Related Medically Attended Visit (MAV) for Management/Treatment of COVID-19 Which May Have Occurred in Any Setting Through Day 29
Description: MAV for management/treatment of COVID-19 may have occurred in any setting e.g., emergency department, urgent care, outpatient clinic, or professional setting wherein direct in-person/telemedicine medical assessment and escalation of care for COVID-19 was provided by licensed healthcare personnel. The percentage of participants requiring at least one COVID-19-related MAV for management/treatment of COVID-19 (apart from routinely scheduled study-directed visits) within each treatment group was presented along with a two-sided exact (Clopper-Pearson) 95% CI.
Time Frame: Up to Day 29
Population: mITT population included the subset of ITT participants who were also dosed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 152 | 153 | 156
percentage of participants | 17.1 [11.5 to 24.0] | 19.0 [13.1 to 26.1] | 14.1 [9.1 to 20.6]
Statistical Analysis 1: Comparison: C19-IG 20% 1 g vs Placebo; Test type: Superiority; p = 0.4676, Chi-squared — p-value was calculated using Chi-square test with 5% level of significance to test the null hypothesis of no difference in the percentage of participants who required at least 1 COVID-19 related MAV between C19-IG 20% 1 g dose group and placebo; Difference in Percentage = 3.0, 95% CI 2-sided [-5.3 to 11.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: C19-IG 20% 2 g vs Placebo; Test type: Superiority; p = 0.2507, Chi-squared — p-value was calculated using Chi-square test with 5% level of significance to test the null hypothesis of no difference in the percentage of participants who required at least 1 COVID-19 related MAV between C19-IG 20% 2 g dose group and placebo; Difference in Percentage = 4.9, 95% CI 2-sided [-3.6 to 13.4] — [estimate comment as in outcome 1, analysis 2]

13. Secondary Outcome: Percentage of Participants Who Required Hospital Admission for Medical Care (Non-Quarantine Purposes) Through Day 29
Description: The percentage of participants requiring hospital admission through Day 29 within each treatment group was presented along with a two-sided exact (Clopper-Pearson) 95% CI.
Time Frame: Up to Day 29
Population: mITT population included the subset of ITT participants who were also dosed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 152 | 153 | 156
percentage of participants | 2.0 [0.4 to 5.7] | 4.6 [1.9 to 9.2] | 1.9 [0.4 to 5.5]
Statistical Analysis 1: Comparison: C19-IG 20% 1 g vs Placebo; Test type: Superiority; p = 0.9744, Chi-squared — p-value was calculated using Chi-square test with 5% level of significance to test the null hypothesis of no difference in the percentage of participants who required hospital admission between C19-IG 20% 1 g dose group and placebo; Difference in Percentage = 0.1, 95% CI 2-sided [-3.8 to 4.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: C19-IG 20% 2 g vs Placebo; Test type: Superiority; p = 0.1878, Chi-squared — p-value was calculated using Chi-square test with 5% level of significance to test the null hypothesis of no difference in the percentage of participants who required hospital admission between C19-IG 20% 2 g dose group and placebo; Difference in Percentage = 2.7, 95% CI 2-sided [-1.6 to 7.5] — [estimate comment as in outcome 1, analysis 2]

14. Secondary Outcome: Duration of Hospital Stay Through Day 29
Description: The duration (number of days) of hospitalization from post-randomization through Day 29 was calculated based on hospital admission and discharge dates recorded.
Time Frame: Up to Day 29
Population: mITT population included the subset of ITT participants who were also dosed. Here, "Overall number of participants analyzed" is the number of participants who were hospitalized.
Measure: Median (Full Range); unit: days
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 3 | 7 | 3
days | 9.0 [6 to 18] | 10.0 [3 to 15] | 9.0 [8 to 15]
Statistical Analysis 1: Comparison: C19-IG 20% 1 g vs Placebo; Test type: Superiority; p = 0.9485, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.38 to 0.40] — 95% CI for difference in LS Mean between C19-IG 20% 1 g dose group and placebo was calculated using ANCOVA model, including length of hospital stay as dependent variable & treatment group as fixed effect, adjusting for baseline
Statistical Analysis 2: Comparison: C19-IG 20% 2 g vs Placebo; Test type: Superiority; p = 0.4734, ANCOVA; LS Mean Difference = 0.14, 95% CI 2-sided [-0.25 to 0.54] — 95% CI for difference in LS Mean between C19-IG 20% 2 g dose group and placebo was calculated using ANCOVA model, including length of hospital stay as dependent variable & treatment group as fixed effect, adjusting for baseline

15. Secondary Outcome: Percentage of Participants Who Required Intensive Care Unit (ICU) Admission or Initiation of ICU Level Care Through Day 29
Description: The percentage of participants requiring ICU admission through Day 29 within each treatment group was presented along with a two-sided exact (Clopper-Pearson) 95% CI. ICU level care is defined as the medical need for intensive or invasive monitoring; the immediate or impending need for the support of the airway, breathing, or circulation; and/or stabilization of acute severe, or life-threatening complications of COVID-19.
Time Frame: Up to Day 29
Population: mITT population included the subset of ITT participants who were also dosed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 152 | 153 | 156
percentage of participants | 0.66 [0.02 to 3.61] | 0.65 [0.02 to 3.59] | 0.64 [0.02 to 3.52]
Statistical Analysis 1: Comparison: C19-IG 20% 1 g vs Placebo; Test type: Superiority; p = 0.9853, Chi-squared — p-value was calculated using Chi-square test with 5% level of significance to test the null hypothesis of no difference in the percentage of participants who required ICU admission between C19-IG 20% 1 g dose group and placebo; Difference in Percentage = 0.02, 95% CI 2-sided [-3.05 to 3.12] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: C19-IG 20% 2 g vs Placebo; Test type: Superiority; p = 0.9890, Chi-squared — p-value was calculated using Chi-square test with 5% level of significance to test the null hypothesis of no difference in the percentage of participants who required ICU admission between C19-IG 20% 2 g dose group and placebo; Difference in Percentage = 0.01, 95% CI 2-sided [-2.99 to 3.07] — [estimate comment as in outcome 1, analysis 2]

16. Secondary Outcome: Duration of ICU Stay Through Day 29
Description: The duration (number of days) of ICU stay from post-randomization through Day 29 was calculated based on ICU admission and discharge dates recorded.
Time Frame: Up to Day 29
Population: mITT population included the subset of ITT participants who were also dosed. Here, "Overall number of participants analyzed" is the number of participants who were admitted to the ICU.
Measure: Median (Full Range); unit: days
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 1 | 1 | 1
days | 7.0 [7 to 7] | 5.0 [5 to 5] | 3.0 [3 to 3]
Statistical Analysis 1: Comparison: C19-IG 20% 1 g vs Placebo; Test type: Superiority; p = 0.5780, ANCOVA; LS Mean Difference = 0.03, 95% CI 2-sided [-0.07 to 0.12] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: C19-IG 20% 2 g vs Placebo; Test type: Superiority; p = 0.9065, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.09 to 0.10] — [estimate comment as in outcome 14, analysis 2]

17. Secondary Outcome: Percentage of Participants Requiring Invasive Mechanical Ventilation Through Day 29
Description: The percentage of participants requiring invasive mechanical ventilation through Day 29 within each treatment group was presented along with a two-sided exact (Clopper-Pearson) 95% CI.
Time Frame: Up to Day 29
Population: mITT population included the subset of ITT participants who were also dosed.
Measure: Number; unit: percentage of participants
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 152 | 153 | 156
percentage of participants | 0.0 | 0.0 | 0.0

18. Secondary Outcome: Duration of Invasive Mechanical Ventilation Through Day 29
Description: The duration (number of days) on invasive mechanical ventilation from post randomization through Day 29 was calculated based on the start/stop dates of invasive mechanical ventilation.
Time Frame: Up to Day 29
Population: No participants required mechanical ventilation throughout the study duration.
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: All-Cause Mortality Through Day 29
Description: All-cause mortality rate is the percentage of participants in each treatment group who experienced mortality up to Day 29.
Time Frame: Up to Day 29
Population: mITT population included the subset of ITT participants who were also dosed.
Measure: Count of Participants; unit: Participants
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 152 | 153 | 156
Participants | 0 | 0 | 0

20. Secondary Outcome: Percentage of Participants With Critical COVID-19 Illness
Description: Critical COVID-19 illness was defined as any one of the following: (a) requiring ICU admission or ICU level of care, (b) invasive mechanical ventilation, or (c) resulting in death by Day 29. The percentage of participants with critical COVID-19 illness defined above within each treatment group was presented along with a two-sided exact (Clopper-Pearson) 95% CI.
Time Frame: Up to Day 29
Population: mITT population included the subset of ITT participants who were also dosed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 152 | 153 | 156
percentage of participants | 0.66 [0.02 to 3.61] | 0.65 [0.02 to 3.59] | 0.64 [0.02 to 3.52]
Statistical Analysis 1: Comparison: C19-IG 20% 1 g vs Placebo; Test type: Superiority; p = 0.9853, Chi-squared — p-value was calculated using Chi-square test with 5% level of significance to test the null hypothesis of no difference in the percentage of participants with critical COVID-19 illness between C19-IG 20% 1 g dose group and placebo; Difference in Percentage = 0.02, 95% CI 2-sided [-3.05 to 3.12] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: C19-IG 20% 2 g vs Placebo; Test type: Superiority; p = 0.9890, Chi-squared — p-value was calculated using Chi-square test with 5% level of significance to test the null hypothesis of no difference in the percentage of participants with critical COVID-19 illness between C19-IG 20% 2 g dose group and placebo; Difference in Percentage = 0.01, 95% CI 2-sided [-2.99 to 3.07] — [estimate comment as in outcome 1, analysis 2]

21. Secondary Outcome: Length of Time to Clinical Progression to Critical COVID-19 Illness Through Day 29
Description: Length of time to clinical progression to critical COVID-19 illness was defined as the time to death, invasive mechanical ventilation, or ICU admission/requiring ICU level of care. ICU level care is defined as the medical need for intensive or invasive monitoring; the immediate or impending need for the support of the airway, breathing, or circulation; and/or stabilization of acute severe, or life-threatening complications of COVID-19. The time to clinical progression was estimated using the KM method.
Time Frame: Up to Day 29
Population: mITT population included the subset of ITT participants who were also dosed. Here, "Overall number of participants analyzed" is the participants who had clinical progression through Day 29. Participants who did not meet the criteria for clinical progression were right censored as of the date of last participant's contact on or prior to Day 29.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 1 | 1 | 1
days | NA [NA to NA] — The median and 95% CI were not estimable due to insufficient number of participants with the events. | NA [NA to NA] — The median and 95% CI were not estimable due to insufficient number of participants with the events. | NA [NA to NA] — The median and 95% CI were not estimable due to insufficient number of participants with the events.

22. Secondary Outcome: Time to COVID-19 Symptoms Through Day 14
Description: Participants were described as symptomatic if they a. experienced at least two of the following systemic symptoms: fever (≥38℃), chills, myalgia, headache, sore throat, cough, fatigue that interferes with activities of daily living, new olfactory/taste disorder(s), and vomiting/diarrhea, b. experienced at least one of the following respiratory signs/symptoms: new or worsening shortness of breath or difficulty breathing, c. experienced a peripheral oxygen saturation by pulse oximetry (SpO2) <94% on room air, or d. had radiographical evidence of pneumonia. Time to COVID-19 symptoms was defined as the time from study drug administration to the first time point when any of the above elements was fulfilled through Day 14. The time to COVID-19 symptoms was estimated using the KM method.
Time Frame: Up to Day 14
Population: mITT population included the subset of ITT participants who were also dosed. Here, "Overall number of participants analyzed" is the number of participants who experienced symptoms through Day 14.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
Number analyzed (Participants) | 61 | 54 | 57
days | NA [NA to NA] — The median and 95% CI were not estimable due to insufficient number of participants with the events. | NA [NA to NA] — The median and 95% CI were not estimable due to insufficient number of participants with the events. | NA [NA to NA] — The median and 95% CI were not estimable due to insufficient number of participants with the events.

ADVERSE EVENTS:
Time Frame: From start of the study up to end of study (up to Day 60)
Description: Safety population included all participants who received any amount of C19-IG 20%/Placebo.
Arm/Group | C19-IG 20% 1 g | C19-IG 20% 2 g | Placebo
All-Cause Mortality (participants affected / at risk) | 0/152 | 0/153 | 0/156
Serious Adverse Events (participants affected / at risk) | 3/152 | 7/153 | 3/156
Other Adverse Events (participants affected / at risk) | 10/152 | 8/153 | 5/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C19-IG 20% 1 g (N=152) | C19-IG 20% 2 g (N=153) | Placebo (N=156)
COVID-19 pneumonia (Infections and infestations) | 3 | 7 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | C19-IG 20% 1 g (N=152) | C19-IG 20% 2 g (N=153) | Placebo (N=156)
Alanine aminotransferase increased (Investigations) | 10 | 8 | 5

LIMITATIONS AND CAVEATS:
The study was terminated for futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT04847141/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT04847141/SAP_001.pdf